CLINICAL TRIAL: NCT05510726
Title: Reliability, Validity, and Responsiveness of Shearwave Elastography to Assess Muscle Stiffness in Neurological Population With Muscle Overacivity
Brief Title: Quantitative Evaluation of Muscle Stiffness in Neurological Patients With Muscle Overactivity
Status: Completed | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/18MAI/217
Record Dates: First submitted 2022-08-17; First posted 2022-08-22 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Muscle Spasticity
Keywords: spasticity; sonoelastography
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: shearwave elastography — shearwave elastography on upper or lower limb

SUMMARY:
Objective:

1. to investigate reliability, validity and responsiveness of shearwave elastography (SWE) to assess muscle stiffness of overactive upper or lower limb muscles in different angle joint positions in patients with neurological condition
2. to investigate the relationship between muscle stiffness measured by SWE and by MyotonPro
3. to investigate the correlation between muscle stiffness measured by SWE and clinical outcomes

Methods: each patient will be assessed three times: two times at an interval of 15 minutes on the same day and one time at an interval of one week at the same time of the day. The following measurements will be made at each evaluation: SWE, MyotonPro, clinical evaluation. SWE and MytotonPro will be taken at different angle joint position.

Outcomes: muscle stiffness measured by SWE and MyotonPro at different angle joint positions, and clinical evaluation (passive range of motion, modified ashworth scale, tardieu scale, fuglmeyer) Hypothesis: SWE is a valid, reliable, and resposive method to assess muscle stiffness in neurological population with muscle overactivity. The results of SWE will be correlated with the results of MyotonPro and with clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* hemiparesia/-plegia following neurological condition (TBI, stroke,...)
* > 3 months after injury
* muscle overactivity in lower limb

Exclusion Criteria:

* other neurological or orthopaedic conditions involving the affected limb
* aphasia or major cognitive impairment limiting functional assessment
* botulinum toxin injection in the last 3 months
* previous treatment of muscle overactivity with surgical procedures.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In- or outpatients of the physical rehabilitation unit of the Cliniques universitaires Saint-Luc
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
reliability, validity and responsiveness shearwave elastography (SWE) to assess muscle elasticity | Day 1
  expressed in m/s. A smaller shearwave velocity indicates a better outcome.
reliability, validity and responsiveness shearwave elastography (SWE) to assess muscle elasticity | Day 1 + 15 minutes
  expressed in m/s. A smaller shearwave velocity indicates a better outcome
reliability, validity and responsiveness shearwave elastography (SWE) to assess muscle elasticity | Day 1 + 7-14 days
  expressed in m/s. A smaller shearwave velocity indicates a better outcome

SECONDARY OUTCOMES:
muscle stiffness assessment with MyotonPro | two times day 1 at 15minutes interval + 7-14 days later at same time of the day
  a smaller muscle stiffness indicates a better outcome

OTHER OUTCOMES:
passive range of motion | day 1 + 7-14 days later at same time of the day
  expressed in angles °. The greater the angle, the better the outcome
modified ashworth scale | day 1 + 7-14 days later at same time of the day
  minimum score:0; maximum score: 4. A higher score indicates a greater spasticity thus a worse outcome
Tardieu scale | day 1 + 7-14 days later at same time of the day
  minimum score:0; maximum score: 4. A higher score indicates a greater spasticity thus a wourse outcome
Fugl-meyer score (Lower extremity; motor function) | day 1 + 7-14 days later at same time of the day
  maximum score of 34. The highest the score, the better the motor function

CONTACTS AND LOCATIONS:
Overall Officials: Gaëtan Stoquart, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No